CLINICAL TRIAL: NCT00083707
Title: UARK 99-006, A Phase II Pilot Study of Anti-Angiogenesis Therapy Using Thalidomide in Patients With Waldenstrom's Macroglobulinemia
Brief Title: Anti-Angiogenesis Therapy Using Thalidomide in Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Celgene Corporation (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 99-006
Record Dates: First submitted 2004-05-27; First posted 2004-05-31 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: Macroglobulinemia; Waldenstrom; Thalidomide
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The purpose of this research is to study how helpful thalidomide is in controlling the disease and to study any side effects from taking thalidomide.

DETAILED DESCRIPTION:
Patients will receive thalidomide in the oral form each night before bed. The dose of thalidomide will be increased each week until week 7 as long as there are no significant side effects.

Routine physical examinations and blood tests will be done to monitor the effect of treatment and the toxicities encountered, if any, and provide the available treatments for side effects accordingly. Blood tests will be done to monitor the tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of previously treated, active Waldenstrom's Macroglobulinemia
* Patients must have adequate hematologic function as demonstrated by total white blood count > or = 2000/mm3, adequate renal function as demonstrated by serum creatinine < or = 3.0 mg/dl, and adequate hepatic function as demonstrated by bilirubin < or = 1.5 mg/dl and transaminases < or = 4 x ULN
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* No other concurrent therapy for WM is permitted while on thalidomide
* Pregnant or nursing women may not participate. Before starting treatment, women of childbearing potential should have a negative pregnancy test performed within 24 hours prior to beginning therapy. Written report of a negative pregnancy test must be obtained before a prescription for thalidomide is issued. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. Pregnancy testing is not required for 1) women who have been post-menopausal for at least 2 years with no menses, 2) women who have had a hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1999-01; Study Completion 2003-02

PRIMARY OUTCOMES:
To determine tumor response, overall and progression free survival following thalidomide therapy in patients with Waldenstrom's Macroglobulinemia (WM)

SECONDARY OUTCOMES:
To determine toxicities associated with thalidomide in patients with Waldenstrom's Macroglobulinemia

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Fassas, M.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu